CLINICAL TRIAL: NCT05268627
Title: Endoscopic Ultrasound Guided Gastric Botulinum Toxin Injections Versus Glucagon Like Peptide 1 Receptor Agonist in Weight Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Asmaa Gameel, principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.21.10.1495
Record Dates: First submitted 2022-01-27; First posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Liraglutide; Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Ultrasound Guided Gastric Botulinum Toxin Injections (Active Comparator)
  Interventions: Drug: Liraglutide
- liraglutide (Active Comparator)
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — endoscopy
  Other Names: Endoscopic ultrasound

SUMMARY:
Background: Obesity is an important public health concern. Surgery is effective but invasive and expensive, and some obese persons are not good surgical candidates.

Aim:

Compare safety, feasibility and efficacy of endoscopic ultrasound guided boutlinum toxin injection and GLP-1 agonists in treatment of obesity.

Methods Full written informed consent will be obtained from all patients.Patient demographics.Detailed medical history.Complete clinical examination.The two methods of intervention will be combined with prescription of several life style modifications as a 2000 kcal diet in men, or 1800kcal in women and moderate daily aerobic exercise (at least 30 minutes, 5 times a week) during 4 months and body weight will be assessed during a 16-week follow-up period.BTA group:Esophagogastroduodenoscopy (EGD) will be done to all subjects under conscious sedation. If no ulceration or retained food, EUS and BTA injection will be performed under the same sedation. EUS examinations will be performed. BTA injections will be made via a 25-gauge EUS needle. A ring of five injections will be made into the gastric antral muscularis propria, 2 to 3 cm proximal to the pylorus. The subjects will receive 20 U at each injection. Subjects will be assessed for complications after recovery from conscious sedation and, again, by telephone the next day.During a 16-week follow-up period after BTA injections, subjects will be weighed weekly.GLP1 group:GLP-1 receptor agonist (Liraglutide subcutaneous once daily).We will start by 0.6 mg daily and we will raise the dose up to 3 mg gradually if patient tolerated.During a 16 week follow up period, subjects will be weighed weekly.

DETAILED DESCRIPTION:
Introduction

Obesity is an important public health concern. Although most pharmacologic therapies have targeted the central nervous system, surgical treatments induce satiation by decreasing the size of the gastric reservoir and inducing maldigestion or malabsorption.

Surgery is effective but invasive and expensive, and some obese persons are not good surgical candidates. Promising pharmacologic and endoscopic approaches to obesity include treatments that affect gastric volume, gastric emptying, gastric compliance, and satiation.

In rats, botulinum toxin A (BTA) injected subserosally into the antrum resulted insignificant decreases in caloric intake and body weight when compared to control and injected rats. Subsequent open-label human studies and three small randomized trials have reported conflicting results, with some studies finding little or no body weight loss after gastric BTA injection and one randomized controlled trial showing statistically significant decreases in gastric emptying and body weight . These trials differed in BTA dose (100 to 300 U in Botox formulation equivalents) and location of injections (antrum alone vs. antrum, body, and cardia). Depth of injection in the gastric wall was largely unknown in these studies, as endoscopic ultrasound (EUS) was not used to guide injection into the muscularis propria or subserosal layers.

In a study by Topazian. (2008), mean body weight reduction was similar in subjects receiving 100 or 300 U BTA (5.0 vs. 4.8 kg). There was a no significant trend toward loss of more body weight in the three subjects who developed decreased gastric emptying after receiving 300 U BTA. Also EUS guidance would help to assure injection of BTA in the gastric muscularis propria and subserosal layers of the gastric wall.

Glucagon-like peptide 1 (GLP-1) is a cleavage product of the pre- proglucagon gene which is expressed in the α-cells of the pancreas, the L-cells of the intestine, and neurons located in the caudal brainstem and hypothalamus. GLP-1 is primarily synthesized and secreted by the L cells of the distal small intestine in response to a nutrient load, although non-nutrient driven secretion has also been reported. GLP-1 is also synthesized by a small population of neurones in the nucleus of the solitary tract (NTS) in the caudal brainstem which project to areas in the hypothalamus and hindbrain that express GLP-1 receptors (GLP-1- R).

In response to a meal, GLP-1 delays gastric emptying and increases gastric volumes. GLP-1 enhances insulin secretion and inhibits glucagon-release in a glucose-dependent manner both in normal individuals as well as in patients with type 2 diabetes. In patients with type 2 diabetes, GLP-1 agonist infusion in pharmacologic doses enhanced satiation and promoted weight loss. Hence GLP-1 therapy in humans reduces food intake, appetite and hunger and promotes fullness and satiety with the ultimate result of promoting weight loss.

The weight loss observed with GLP-1 agonist therapy may be associated with reductions in total body fat, in particular visceral and truncal adipose.

Also of interest is the successful use of GLP-1 agonists in the treatment of hypothalamic obesity, suggesting that at least in this cohort, GLP-1 analogues were capable of inducing weight loss despite hypothalamic damage.

Unlike pure dietary measures, weight loss may be sustained for up to a period of 3 years in the presence of GLP-1 agonist therapy. However, once therapy is discontinued, there is some regain of weight. There seems to be minimal effect of GLP-1 on energy expenditure per se and thus the overall negative energy balance seen with GLP-1 therapy is largely a result of decreased energy intake.

Aim of work Compare safety, feasibility and efficacy of endoscopic ultrasound guided boutlinum toxin injection and GLP-1 agonists in treatment of obesity.

Patients and Methods Patients Study Design Prospective randomized study.

Study groups 2 Groups: First one: BTA will be injected into gastric antral muscularis propria under EUS guidance.

Second group: will receive GLP-1 receptor agonist (Liraglutide subcutaneous once daily) Methods

1. Full written informed consent will be obtained from all patients.
2. Patient demographics.
3. Detailed medical history
4. Complete clinical examination
5. The two methods of intervention will be combined with prescription of several life style modifications as a 2000 kcal diet in men, or 1800kcal in women and moderate daily aerobic exercise (at least 30 minutes, 5 times a week) during 4 months and body weight will be assessed during a 16-week follow-up period.
6. BTA group Esophagogastroduodenoscopy (EGD) will be done to all subjects under conscious sedation. If no ulceration or retained food, EUS and BTA injection will be performed under the same sedation. EUS examinations will be performed. BTA injections will be made via a 25-gauge EUS needle. A ring of five injections will be made into the gastric antral muscularis propria, 2 to 3 cm proximal to the pylorus. The subjects will receive 20 U at each injection. Subjects will be assessed for complications after recovery from conscious sedation and, again, by telephone the next day.During a 16-week follow-up period after BTA injections, subjects will be weighed weekly.
7. GLP1 group GLP-1 receptor agonist (Liraglutide subcutaneous once daily).the investigators will start by 0.6 mg daily and raise the dose up to 3 mg gradually if patient tolerated.During a 16 week follow up period, subjects will be weighed weekly.

ELIGIBILITY:
Inclusion Criteria:

Sex: both Age: from 20 to 60 years Body Mass Index > 30

Exclusion Criteria:

Age: below 20 or above 60 years old. Patient with known gastroparesis Peptic ulcer disease or active upper gastrointestinal ulceration Prior gastric or small bowel surgery American Society of Anesthesiologists (ASA) class 3 or higher Patients with more than mild , infrequent symptoms of upper abdominal pain or nausea Pregnant or lactating female Contraindications of sedation (Uncontrolled Diabetes Mellitus, Uncontrolled Thyroid Disorders, Pregnancy, Respiratory Embarrassment, Reactional Drugs like Antidepressants and Anti-anxiety Agents).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-01-27 (Estimated); Study Completion 2023-01-27 (Estimated)

PRIMARY OUTCOMES:
weight loss | 1 year
  weight in kilograms
Body mass index | 1 year
  BMI weight/ height2
waist circumference | 1 year
  waist circumference in cm
hip circumference | 1 year
  hip circumference in cm

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Specialized Medical Hospital,Mansoura University, Al Mansurah, Dakhlia
  - MansouraU, Al Mansurah

IPD SHARING:
Plan to Share IPD: Undecided